CLINICAL TRIAL: NCT02356497
Title: Prospective Evaluation of Interventional Studies on Bone Metastases - the PRESENT Cohort
Acronym: PRESENT
Status: Recruiting | Type: Observational
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Helena M Verkooijen, Prof. dr., UMC Utrecht
Other Study IDs: NL49273.041.14
Record Dates: First submitted 2015-02-01; First posted 2015-02-05 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Bone Metastases
Keywords: Bone metastases; Metastatic bone disease; Multi-trial facility
MeSH Terms: conditions — Bone Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Bone metastases are frequent distant manifestations of cancer, with pain as a common and devastating consequence. The primary treatment for painful bone metastases, external beam radiation therapy, is moderately effective: about 60% of patients who undergo conventional radiotherapy experience (partial) pain relief. Several factors associated with treatment failure have been identified, but no attempts have been made to collapse these factors into a clinically useful prediction tool to predict treatment response. In addition, to aid in therapy selection based on expected survival time, development of survival models is essential. Finally, we need innovative treatments as alternatives or additive to standard treatment options to improve quality of life (QoL). For these reasons, we set up the PRESENT cohort study, recruiting patients at the departments of radiation oncology and orthopedic surgery.

We aim to provide detailed information about clinical data, create an infrastructure for efficient, fast and pragmatic evaluation and implementation of innovative interventions, as well as development of accurate new prediction tools.

DETAILED DESCRIPTION:
The PRESENT cohort is set up according to the 'cohort multiple Randomised Controlled Trial' design. The basis of this design is a prospective cohort of patients with bone metastases, receiving care as usual, who give informed consent for cohort participation. At the UMC Utrecht, patients are furthermore asked for informed consent to be randomized in future RCTs conducted within the cohort. Patients are informed that they will be offered the experimental intervention if they are randomly selected. They are also informed that they otherwise might serve as controls without being notified and that their data can be used in a trial context. For each patient in the cohort, clinical and patient-reported outcomes are captured at baseline and at regular intervals during follow-up. Within this cohort, multiple RCTs can be conducted. For this purpose, eligible patients who have provided the consent required for them to participate in an RCT within the cohort are identified. From this subcohort, a random selection of patients will be invited to undergo the experimental intervention. Eligible participants who were not randomly selected receive standard care, are not informed about the experimental intervention and serve as controls. Outcomes in this control group are compared with the outcomes of those who were offered the experimental intervention, in order to estimate the effect of the experimental intervention versus usual care. Within the cohort, the same process can be repeated for trials of other interventions.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of malignancy;
* Radiographic or histologic proof of metastatic bone disease;
* Undergoing radiotherapy;
* Age > 18 years;
* Informed consent - at least - for use of routinely collected clinical data.

Exclusion Criteria:

* Mentally incompetent patients;
* Life expectancy < 1 week indicated by the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with bone metastases undergoing radiotherapy will be asked to participate in this cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2013-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pain response | at 2, 4, 6, 8 weeks, 3 and 6 months, then every 6 months

SECONDARY OUTCOMES:
Health-related Quality of Life | at 2, 4, 6, 8 weeks and 3 months
Toxicity according to CTCAE version 4 | up to 3 months
  Grade 3 and 4 side effects occurring during or up to 3 months after radiotherapy will be registered according to the Common Terminology Criteria for Adverse Events (CTCAE version 4). The following side effects will be registered: Nausea; Vomiting; Diarrhoea; Pain flare.
Readmission | up to 3 years
  Reintervention (reirradiation, surgery, other); Development of neurological symptoms; Development of pathologic fracture
Survival | up to 3 years
  Survival of participating patients will be recorded using the follow up questionnaires (returned by family members) or are derived from the Municipal Personal Records Database (in Dutch: Gemeentelijke Basisadministratie, GBA).

CONTACTS AND LOCATIONS:
Overall Officials: Helena M. Verkooijen, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Current enrolment approaches 2000 patients. Investigators are encouraged to request data after consulting the study team.

REFERENCES:
- See also: Related Info — http://www.radiotherapie.nl/